CLINICAL TRIAL: NCT03968133
Title: Treating Anxiety in Parkinson's Disease With a Multi-Strain Probiotic - a Randomized, Placebo-controlled Trial
Brief Title: Treating Anxiety in Parkinson's Disease With a Multi-Strain Probiotic
Acronym: TAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: The W. Garfield Weston Foundation (Unknown)
Responsible Party: Principal Investigator, Silke Cresswell, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H18-03083
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease; Anxiety
Keywords: probiotic; mood
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized, triple-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Ecologic® BARRIER 849 (Maize starch, maltodextrin, vegetable protein, potassium chloride, +/- probiotic bacteria (B. bifidum W23, B. lactis W51, B. lactis W52, L. acidophilus W37, L. brevis W63, L. casei W56, L. salivarius W24, Lc. lactis W19, Lc. lactis W58; ≥ 2,5*10^9 colony forming unit (CFU)/g), magnesium sulphate, manganese sulphate.) sachet, two times daily dosing for a total of 2 grams (viable cell count of 2.5 × 10^9 CFU/gram) per day.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo (maize starch, maltodextrin, vegetable protein, magnesium sulphate, manganese sulphate)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Oral probiotic delivered in powdered form.
  Other Names: Ecologic® BARRIER 849
  Arms: Probiotic
Dietary Supplement: Placebo — Oral placebo delivered in powdered form.
  Arms: Placebo

SUMMARY:
This study evaluates the use of an oral multi-strain probiotic in the treatment of anxiety in individuals with Parkinson's Disease. Participants will be randomized to either 12-week multi-strain probiotic treatment or placebo.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a complex condition that carries a high burden of neuropsychiatric comorbidities. About a third of individuals living with Parkinson's disease have one or more anxiety disorders, resulting in lower quality of life, greater care dependency, and increased caregiver burden. Gastrointestinal dysfunction is very common in Parkinson's. Constipation is experienced by the vast majority of patients and often manifests years before onset of motor symptoms, symptoms suggestive of irritable bowel syndrome are also commonly found in PD. Increased intestinal permeability has been demonstrated in PD. Impaired intestinal barrier function can lead to chronic systemic low-grade inflammation, which has been strongly associated with mood disorders. Several lines of evidence suggest a link between the gut microbiome and Parkinson's disease.

The microbiome has been linked to anxiety both in human and animal studies. Several studies have found beneficial effects of probiotics on mood disorders in non-PD populations, including stress and depressive behaviour in animal models, and sad mood reactivity and major depressive disorder in humans. Specifically regarding anxiety, probiotics have shown benefits in several animal models; human probiotic trials have demonstrated improvements in psychological distress and anxiety in healthy controls, in mothers experiencing postpartum depression and anxiety and in individuals afflicted with IBS-related anxiety without PD.

In summary, given the high rate of anxiety in PD, the growing evidence that probiotics may improve anxiety and mood disorders in non-PD populations, and the strong links between the gut microbiome and PD, we will carry out a randomized, blinded, placebo-controlled study into the use of a multi-strain probiotic to improve anxiety and Parkinson's disease.

Recruitment: Approximately 72 participants will be randomized to either the probiotic intervention arm or placebo treatment. Participants will mainly be recruited from the Pacific Parkinson's Research Centre movement disorder clinic at the University of British Columbia in Vancouver.

Participants will receive a detailed description of the study and will need to provide informed consent for participation in the study. Participants will be screened for inclusion and exclusion criteria.

Assessments: Clinical assessments of motor function, cognition and neuropsychiatric symptoms will be done before the 12 week intervention phase as well as following after the 12 week intervention with regular check ins during the course of the intervention. Blood samples and stool samples will be collected before and after the intervention.

The primary outcome will be the difference between the probiotic vs. placebo groups in mean Parkinson's Anxiety Scale (PAS) score pre/post-intervention. The primary analysis will be based on intention-to-treat. Secondary analyses for anxiety will include assessing the proportion of participants with a post-intervention PAS of ≤13 in each group. For other secondary outcomes, the between-group difference analysis will be applied to the fatigue, depression, PD motor function, severity (UPDRS I-III) and quality of life scores pre/post intervention, respectively. Adverse events, tolerability and drop-out rates will be registered and overall rates compared between the intervention groups. Furthermore, differences and changes in blood markers and microbiome composition will be assessed.

ELIGIBILITY:
Inclusion Criteria

1. Confirmed diagnosis of Parkinson's disease based on Queen Square Brain Bank criteria
2. Between ages 40-80
3. Hoehn and Yahr stage between 1-3 (mild to moderate PD) in the "ON" state
4. Anxiety (PAS score ≥14, MDS-UPDRS Part 1.4 score ≥ 2, and/or clinical diagnosis of anxiety based on the MINI clinical interview in the "ON" state)
5. Women of childbearing potential must agree to use a medically approved method of birth control (e.g. hormonal contraceptives, intrauterine devices, vasectomy/tubal litigation, barrier methods and double barrier method) and must have a negative urine pregnancy test result at screening and baseline
6. Willingness to maintain current physical activity levels during study period

Exclusion criteria

1. Atypical parkinsonism
2. Active suicidality
3. Active psychosis
4. Cognitive score (MoCA) of <21 in "ON" state
5. BDI-II score above 28 in "ON" state
6. Probiotic, sacchromyces boulardii and/or antibiotic usage in the past 3 months
7. Anti-inflammatory drug usage more than twice a week (e.g. corticosteroids, naproxen, ibuprofen, celecoxib). Use of daily 81 mg ASA permitted
8. The use of natural health products that affect depression (e.g. St. John's Wort, passion flower)
9. Concurrent psychotherapy or brain stimulation for the treatment of mood disorders
10. Change in antidepressant or anxiolytic medication (including benzodiazepines) within the last 4 weeks
11. Change in Parkinson's medication within the last 2 weeks
12. Neurological disease other than PD, including Alzheimer's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, a brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma
13. An immune-compromised condition (e.g. AIDS, lymphoma, patients undergoing long term corticosteroid treatment)
14. A bleeding disorder
15. Current illness (for example a cold or flu like symptoms) and infections (for example hepatitis, HIV, gastroenteritis, fungal, or parasitic infections)
16. Allergy to corn starch or corn
17. Concurrent treatment for Parkinson Disease with Duodopa or Deep Brain Stimulation (DBS)
18. Women who are pregnant, breast feeding, or planning to become pregnant during the course of the trial
19. Unstable medical conditions or serious disease/conditions (e.g. cancer, cardiovascular, renal, lung, diabetes)
20. Drug and/or substance abuse

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Parkinson's Anxiety Scale (PAS) | 13 weeks
  The PAS is a self reported 12-item scale that has three subscales: persistent anxiety, episodic anxiety, and avoidance behavior; It is rated using a Likert scale (0-4).

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | 13 weeks
  The BDI is a self reported 21-question multiple-choice self-report inventory on a scale from 0-3.
Parkinson's Disease Quality of Life Questionnaire (PDQ-39) | 13 weeks
  The PDQ-39 is a self reported questionnaire that assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living.
Fatigue Severity Scale (FSS) | 13 weeks
  The Fatigue Severity Scale is a self reported 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders on a scale from 1 (strongly disagree) to 7 (strongly agree).
Montreal Cognitive Assessment | 13 weeks
  The MoCA test is a one-page 30-point administered assessment used for detecting cognitive impairment.
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 13 weeks
  The MDS-UPDRS is a clinical assessment of motor and non-motor symptoms in individuals with Parkinson's Disease. It consists of four subscales. Subscales 1, 3, and 4 are administered by a trained individual with subscale 2 being self reported. Each item is rated from 0 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Silke Appel-Cresswell, MD, Principal Investigator — University of British Columbia
Locations (1):
- Pacific Parkinson's Research Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Lam JS, Tosefsky KN, Zhu J, Meng D, Uzelman P, Pio F, Ainsworth NJ, Vila-Rodriguez F, Howard AK, Appel-Cresswell S. Anxiety is associated with increased risk of suicidality in Parkinson's disease. J Parkinsons Dis. 2026 Jan 6:1877718X251410887. doi: 10.1177/1877718X251410887. Online ahead of print. PMID 41493876